CLINICAL TRIAL: NCT00987311
Title: Pilot Study on the Effects of Probiotic Fermented Dairy Drinks on the Intestinal Immune Response in Healthy Adults
Brief Title: Effect of Probiotic Fermented Dairy Drinks on Intestinal Immune Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NU311
Record Dates: First submitted 2009-09-28; First posted 2009-09-30 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
Keywords: Probiotics; intestinal immune system; human; healthy subjects; dairy drink; Healthy adults
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1-Test product A (Active Comparator): 1-Dairy product containing probiotics A (test product A)
  Interventions: Dietary Supplement: 1- Dairy drink containing probiotics A
- 2-Test product B (Active Comparator): 2-Dairy product containing probiotics B (test product B)
  Interventions: Dietary Supplement: 2- Dairy drink containing probiotics B
- 3-Control (Sham Comparator): 3-Dairy product without probiotics (control)
  Interventions: Dietary Supplement: 3- Dairy drink without probiotics (control)

INTERVENTIONS:
Dietary Supplement: 1- Dairy drink containing probiotics A — 1- Dairy drink containing probiotics A
  Arms: 1-Test product A
Dietary Supplement: 2- Dairy drink containing probiotics B — 2- Dairy drink containing probiotics B
  Arms: 2-Test product B
Dietary Supplement: 3- Dairy drink without probiotics (control) — 3- Dairy drink without probiotics (control)
  Arms: 3-Control

SUMMARY:
The purpose of this study is to investigate whether two different fermented dairy drinks consumed daily could have an effect on the intestinal immune response in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male/female subjects aged from 18 to 45 years (bounds included).
* Subjects with none of the symptoms of gastrointestinal infectious diseases
* Subjects with a body mass index (BMI) between 19 and 30 kg/m² (bounds included).
* Subjects who accept to be submitted to an alimentary restriction of product with OTC and foods containing probiotics and/or prebiotics
* Subjects who regularly consume and appreciate dairy products
* Subjects who have not consumed any products or OTCs containing probiotics within the last three months.

Exclusion Criteria:

* Subjects in a situation that, in the investigator opinion, could interfere with optimal participation in the present study (e.g. non dairy-products consumer) or could constitute a special risk for the subject.
* Subjects with allergies or hypersensitivity to any component of the study product (e.g: allergy or hypersensitivity to milk proteins, or lactose intolerance)
* Subjects with any food allergy
* Subjects with auto-immune or with chronic disease or with a history of chronic metabolic or gastrointestinal.
* Subjects who have had any surgery or intervention requiring general anaesthesia in the last 4 weeks..
* Subjects with special diet requirements
* For female subjects: pregnancy, breast feeding or no method of contraceptive used
* Subjects participating in any other interventional study concomitantly or within 4 weeks of the study entry date.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2011-12 (Actual)